CLINICAL TRIAL: NCT00440778
Title: A Randomized Trial of Early Discharge After Trans-radial Stenting of Coronary Arteries in Acute Myocardial Infarction: The EASY-MI Pilot Study.
Brief Title: A Randomized Trial of Early Discharge After Trans-radial Stenting of Coronary Arteries in Acute MI
Acronym: EASY-MI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Eli Lilly and Company (Industry); Cordis US Corp. (Industry); Quebec Heart Institute (Other)
Responsible Party: Principal Investigator, Olivier F. Bertrand, MD, PhD, Laval University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EASY-MI
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Myocardial Infarction; Ischemia
Keywords: Coronary artery stenting; Trans-radial; Intracoronary
MeSH Terms: conditions — Myocardial Infarction; Ischemia | interventions — Abciximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Gr 1 - intracoronary + infusion (Experimental): abciximab bolus 0.25 mg/kg ic + 12 hrs iv infusion
  Interventions: Drug: Abciximab
- Gr 2 - intracoronary (Experimental): 100% abciximab bolus dose 0.3 mg/kg ic
  Interventions: Drug: Abciximab
- Gr 3 - intravenous (Active Comparator): abciximab bolus dose 0.25 mg/kg iv + 12 hrs iv infusion
  Interventions: Drug: Abciximab
- Gr 4 - intravenous (Experimental): 100% abciximab bolus dose 0.3 mg/kg iv
  Interventions: Drug: Abciximab

INTERVENTIONS:
Drug: Abciximab — 100% abciximab bolus dose (0.3 mg/kg) ic or iv vs standard bolus (0.25 mg/kg) ic or iv plus 12-hr infusion
  Other Names: Abciximab (ReoPro)

SUMMARY:
HYPOTHESES

1. Bolus administration of total abciximab dose provides superior maximal and mean platelet aggregation inhibition (PAI) compared with standard bolus (0.25 mg/kg) administration.
2. Total dose of abciximab can be given as a single bolus and is more effective than bolus (0.25 mg/kg) + 12 hrs infusion in terms of acute and mid-term angiographic and clinical results.
3. Intracoronary (ic) abciximab administration is more effective than intravenous (iv) route of administration in terms of acute and mid-term angiographic and clinical results.
4. There is a relationship between PAI and angiographic perfusion scores.
5. Routine use of sirolimus-eluting stents (Cypher, Cordis) in primary-PCI is associated with a low rate of target vessel revascularization and complications.
6. Cardiac MRI early and late after primary-PCI provides detailed information on myocardial injury and irreversible necrosis, which are correlated with angiographic perfusion scores.
7. After uncomplicated trans-radial PCI, patients can be retransferred early to their referring center.

DETAILED DESCRIPTION:
OBJECTIVES AND END-POINTS The objectives of the present study are to assess the benefits and safety of 1) a single bolus of abciximab (100% dose) compared with the standard bolus (ca 80% of the total dose) + 12h infusion (ca 20% of the total dose), and 2) intracoronary abciximab bolus administration compared with intravenous route of abciximab administration in primary PCI.

The primary PLATELETS end-points are the percentage of patients with ≥ 95% platelet aggregation inhibition 10 minutes after abciximab bolus (MAX) and the mean platelet aggregation inhibition 10 minutes after abciximab bolus (MEAN).

The secondary CLINICAL end-points of the study are:

* The composite of death, stroke, repeat myocardial infarction, urgent target vessel revascularization and major bleedings at 30 days following primary PCI.
* The composite of cardiovascular death, repeat myocardial infarction and repeat target vessel revascularization at 6-months follow-up.

The secondary ANGIOGRAPHIC end-points of the study are:

* The proportion of patients having myocardial blush grade 2-3 and TIMI 3 score at the end of PCI in the culprit vessel.
* The restenosis rate (diameter stenosis ≥ 50%) and late loss in the culprit vessel at 6-months follow-up.

Other exploratory end-points are the feasibility and safety of early transfer to the referring hospital after uncomplicated primary PCI, the cardiac MRI measurements and platelet aggregation inhibition at 6h post-PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute myocardial infarction eligible for primary PCI within 6 h of symptoms: patient must have prolonged, continuous (lasting at least 20 minutes) signs and symptoms of ischemia not eliminated with nitrates and onset within 6 h of randomization, and one of the following:

  * ST-segment elevation ≥ 2 mm in 2 or more contiguous precordial ECG leads (anterior infarction)
  * ST-segment depression ≥ 2 mm in V1, V2 or V2, V3 with reciprocal 1 mm ST-elevation in II, augmented unipolar foot (left leg) lead (AVF), and V6 (true posterior infarction)
  * ST-segment elevation ≥ 1 mm in 2 or more contiguous limb ECG leads (other infarction)
  * New or presumably new left bundle branch block (LBBB)
* Patient must be > 18 years of age.
* Patient and treating interventional cardiologist agree for randomization.
* Patient will be informed of the randomization process and will sign an informed consent.
* Diagnostic and therapeutic intervention performed through trans-radial/ulnar artery approach.
* The culprit lesion can be identified on a native coronary vessel, which is suitable for primary PCI with stent implantation.

Exclusion Criteria:

* Patient has received thrombolytic therapy (within the last 4 weeks) and is referred for rescue PCI
* Concurrent participation in other investigational study
* Femoral sheath (artery)
* Intolerance or allergy to ASA, clopidogrel or ticlopidine precluding treatment for at least 12 months
* Any significant blood dyscrasia, diathesis or INR > 2.0
* Any clinical contraindication to abciximab (ReoPro®) administration i.e. known structural intracranial lesion, thrombocytopenia < 100,000, active or recent bleeding or hemoglobin level known < 10 g/dl.
* Any glycoprotein IIb-IIIa inhibitors use in the previous 30 days
* Uncontrolled high blood pressure i.e. systolic blood pressure ≥ 180 mmHg and/or diastolic blood pressure ≥ 100 mmHg.
* Life expectancy less than 6 months owing to non-cardiac cause
* Infarction caused by in-stent thrombosis or restenosis
* Cardiogenic shock evident before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with at least 95% platelet aggregation inhibition, and mean platelet aggregation inhibition. | 10 min after bolus of abciximab

SECONDARY OUTCOMES:
Composite of death, stroke, repeat MI, urgent target vessel revascularization and major bleedings at 30 days following primary PCI. | 30 days
Composite of cardiovascular death, repeat MI and repeat target vessel revascularization at 6-month follow-up. | 6 months
Proportion of patients having myocardial blush grade 2-3 and TIMI 3 score at the end of PCI in the culprit vessel. | At end of PCI
Restenosis rate (diameter stenosis equal or higher than 50%) and late loss in the culprit vessel at 6-month follow-up. | 6 months
Exploratory end-points: feasibility and safety of early transfer to the referring hospital after uncomplicated primary PCI, cardiac MRI measurements and platelet aggregation inhibition at 6hr post-PCI. | At 6hr post-PCI

CONTACTS AND LOCATIONS:
Overall Officials: Olivier F Bertrand, MD, PhD, Principal Investigator — Laval Hospital Research Center
Locations (1):
- Laval Hospital, Québec, Quebec, Canada

REFERENCES:
- [Derived] Bertrand OF, Larose E, Costerousse O, Mongrain R, Rodes-Cabau J, Dery JP, Nguyen CM, Barbeau G, Gleeton O, Proulx G, De Larochelliere R, Noel B, Roy L. Effects of aspiration thrombectomy on necrosis size and ejection fraction after transradial percutaneous coronary intervention in acute ST-elevation myocardial infarction. Catheter Cardiovasc Interv. 2011 Mar 1;77(4):475-82. doi: 10.1002/ccd.22692. PMID 20578162